CLINICAL TRIAL: NCT05340868
Title: Genetics of the Acute Response to Oral Semaglutide (GAROS)
Brief Title: Genetics of the Acute Response to Oral Semaglutide
Acronym: GAROS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APK.002.12.2022
Record Dates: First submitted 2022-04-01; First posted 2022-04-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-11

CONDITIONS: PreDiabetes; Prediabetic State; Obesity
Keywords: pharmacogenetics; semaglutide; prediabetes; obesity
MeSH Terms: conditions — Prediabetic State; Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Semaglutide (oral) (Experimental): In this study, each participant will receive a regimen of oral semaglutide, a glucagon-like peptide-1 (GLP-1) receptor agonist, for a duration of twelve weeks. The dosage will begin at 3 mg/day for weeks 1-2, gradually increasing to 7 mg/day for weeks 3-4, 14 mg/day for weeks 5-6, 28 mg/day for weeks 7-8, and finally, to 42 mg/day for the last four weeks (weeks 9-12).
  Interventions: Drug: Semaglutide Pill

INTERVENTIONS:
Drug: Semaglutide Pill — Oral semaglutide treatment
  Other Names: Rybelsus

SUMMARY:
The study aims to investigate the genetic basis of the response to short-term (3 months) orally administered semaglutide treatment, in terms of improving metabolic parameters, including the hormonal response to a standardized meal, and changes in body composition and liver steatosis. In the study, parameters such as fasting and 2-hour glucose during OGTT, HbA1c, body fat mass, body weight, total cholesterol, HDL and LDL, triglycerides, HOMA-IR, Matsuda Index and liver steatosis will be assessed. All the patients will undergo genome-wide genotyping. Moreover, in a subset of participants, muscle and fat biopsies will be performed, before and after the treatment, and liver, muscle and pancreas fat content will be assessed using MRI.

DETAILED DESCRIPTION:
Each subject will participate in the following visits:

Visit v1 (screening) - for each patient, fasting venous blood will be collected and an oral glucose tolerance test (OGTT) will be performed - with blood samples taken 30, 60, 90 and 120 minutes after drinking the glucose solution. Fasting blood samples will be used to measure basic metabolic parameters (including glucose, lipid profile, HbA1c, AST, ALT, GGTP, electrolytes, blood count, the presence of antibodies against beta-cell antigens, TSH), and from blood collected at each time point during the OGTT glucose and insulin concentrations will be measured. Each patient will also undergo a detailed body composition analysis using bioimpedance and DXA. In addition, during the visit, each participant will receive a continuous glucose monitoring system (CGM) and an accelerometer to measure physical activity for a period of 10-14 days.

Visit v2 (14-30 days after v1)- during the visit, each patient will undergo a mixed meal tolerance test (MMTT), with blood samples taken 5, 10, 15, 30, 60, 90, 120, 180 minutes after eating the meal, along with a non-invasive measurement of resting energy expenditure (RMR). After the end of the test, the patient will receive semaglutide in two marked doses: 3 mg and 7 mg, along with instructions on how to take them and a diary in which the drug intake and occurrence of side effects will be recorded.

Visit v3 - four weeks after starting the semaglutide treatment. During the visit, fasting venous blood will be collected to measure basic metabolic parameters. Each patient will undergo a detailed body composition analysis using bioimpedance and DXA. During the visit, patients will receive semaglutide in the dose of 14 mg, along with instructions on how to take them and a diary in which the drug intake and occurrence of side effects will be recorded.

Visit v4 - twelve weeks after starting semaglutide treatment. Similar to visit 1 (OGTT).

Visit v5 - twelve weeks after starting semaglutide treatment. Similar to visit 2 (MMTT).

Visit v6 (follow-up visit) - after twelve weeks of ending the semaglutide treatment. Similar to visit 1 (OGTT).

Additionally, a random 20% of the study group will participate in additional visits:

Visit A.1 (between visits v1 and v2), A.2 (+ 1-5 days from visit v5) and A.3 (+ 1-5 days from visit v6) - during the visit, biological material will be collected for each patient in the form of a biopsy of the vastus lateralis muscle and subcutaneous adipose tissue.

Visit B.1 (between visits v1 and v2), B.2 (+ 1-5 days from visit v5) and B.3 (+ 1-5 days from visit v6)- during the visit, patients will undergo an abdominal MRI scan to assess the steatosis of the liver, muscle and pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent was given before any study-related action on the subject.
* Age: 18-65 years old
* Body mass index (BMI) >30 kg/m2 or >27 kg/m2 when accompanied by prediabetes, diagnosed according to the criteria of the American Diabetes Association

Exclusion Criteria:

* Patients diagnosed with a serious chronic disease, including:

  * Ischemic heart disease
  * Heart failure (NYHA class III-IV)
  * Severe renal insufficiency (eGFR <30 ml/min)
  * Severe liver diseases
  * Inflammatory bowel disease
  * Diabetic gastroparesis
  * Cancer - currently or in the last five years prior to screening
  * Chronic obstructive pulmonary disease
  * History of mental illness, major depression or other severe mental disorders
* Use of any medications with clinically-proven significant weight gain or loss effects
* History of undergoing bariatric surgery or other surgery involving the stomach that could affect the absorption of the study drug (according to the investigator's opinion)
* History of idiopathic acute pancreatitis
* A family or personal history of multiple endocrine neoplasia type 2 (MEN2) or medullary thyroid cancer
* For women - pregnancy, breastfeeding or planning pregnancy.
* Women of childbearing age who are not using highly effective methods of contraception
* Known or suspected hypersensitivity to the test product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic measures - change in HbA1c (%) | 1 and 3 months
  Investigators will measure the change in HbA1c concentration between Visit 2, Visit 3 and Visit 4 as an index of Semaglutide response, and compare them by genotype at selected loci.
Body composition - change in body weight (kg) | 1 and 3 months
  Investigators will measure the change in body weight measures between Visit 2, Visit 3 and Visit 4 as an index of Semaglutide response, and compare them by genotype at selected loci.

SECONDARY OUTCOMES:
Glycemic measures - change in 2-hour glucose (in mg/dl) | 1 and 3 months
  Investigators will measure the change in 2-hour glucose measures (OGTT) between Visit 2, Visit 3 and Visit 4 as an index of Semaglutide response, and compare them by genotype at selected loci.
Glycemic measures - change in fasting glucose (in mg/dl) | 1 and 3 months
  Investigators will measure the change in fasting glucose measures between Visit 2, Visit 3 and Visit 4 as an index of Semaglutide response, and compare them by genotype at selected loci.
Body composition - change in body fat content (kg) | 1 and 3 months
  Investigators will measure the change in body fat content between Visit 2, Visit 3 and Visit 4 as an index of Semaglutide response, and compare them by genotype at selected loci.
Body composition - change in lean body mass content (kg) | 1 and 3 months
  Investigators will measure the change in lean body mass content between Visit 2, Visit 3 and Visit 4 as an index of Semaglutide response, and compare them by genotype at selected loci.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szczerbinski, MD, PhD, Principal Investigator — Clinical Research Centre, Medical University of Bialystok
Locations (1):
- Clinical Research Centre, Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in pharmacogenomics. Data or samples shared will be coded, with no PHI included.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
URL: http://umb.edu.pl